CLINICAL TRIAL: NCT01242813
Title: An Open-label, Multicenter, Efficacy and Safety Study of 4-month Canakinumab Treatment With 6-month Follow-up in Patients With Active Recurrent or Chronic TNF-receptor Associated Periodic Syndrome (TRAPS).
Brief Title: Efficacy and Safety Study of ACZ885 in Patients With Active Recurrent or Chronic TNF-receptor Associated Periodic Syndrome (TRAPS).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2203; 2010-020061-24
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: TNF-receptor Associated Periodic Syndromes (TRAPS)
Keywords: TNF-receptor associated periodic syndrome; fevers; rashes; musculoskeletal and abdominal pain; periorbital edema; TNFR1
MeSH Terms: conditions — Periodic fever, familial, autosomal dominant; Fever; Exanthema; Abdominal Pain; Orbital Cellulitis | interventions — canakinumab

ARMS (1):
- Canakinumab (Experimental): This was an open-label, single treatment arm, multicenter study of monthly canakinumab 150 mg (2 mg/kg for patient ≤ 40 kg) subcutaneous injections in patients with active recurrent or chronic TRAPS.
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885

SUMMARY:
This trial will assess the safety and efficacy of ACZ885 in patients with active recurrent or chronic TNF-receptor associated periodic syndrome (TRAPS).

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent for >or= 18 years of age before any assessment is performed. Parent or legal guardian's written informed consent and child's assent, if appropriate, are required before any assessment is performed for patients < 18 years of age.
2. Male and female patients at least 4 years of age at the time of the screening visit.
3. Patients with a clinical diagnosis of TRAPS and a mutation of TNFRSF1A gene. Patients with low penetrance mutations, such as R92Q or P46L, can be included with mutual agreement between the investigator and Novartis.
4. Patients with a diagnosis of recurrent TRAPS must experience more than 6 episodes/year prior to receiving an effective biologic therapy and the duration of each episode lasted at least 8 days. For patients receiving biologic therapy, this criterion applies to prior to receiving the biologic therapy.
5. Patients who have been treated with anakinra must have demonstrated a partial or complete clinical response with an associated decrease in their inflammation markers (CRP and SAA).
6. Active TRAPS as evidenced by clinical signs and symptoms of active TRAPS (Physician's Global Assessment >or= 2) and an elevated CRP > 10mg/L (Normal CRP range <or= 10 mg/L) and/or SAA > 10 mg/L (Normal SAA range <or= 10 mg/L) at time of first canakinumab treatment.

Exclusion Criteria:

1. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
2. Women of child-bearing potential, defined as pre-menarche females aged 8 years and above or all women physiologically capable of becoming pregnant, UNLESS they are

   * women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner
   * women whose partners have been sterilized by vasectomy or other means
   * using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices [IUDs]; periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] is not acceptable) or total abstinence at the discretion of the investigator in cases where the age, career, lifestyle, or sexual orientation of the patient ensures compliance.
   * Women of child-bearing potential should be willing to use a reliable contraception throughout the study and for 3 months after study drug discontinuation.
   * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
3. History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot) test result.
4. Positive QuantiFERON (QFT-TB G In-Tube) test or positive Purified Protein Derivative (PPD) test (>or= 5 mm induration) at screening or within 2 month prior to the screening visit, according to the national guidelines. Patients with a positive PPD test (>or= 5 mm induration) at screening may be enrolled only if they have either a negative chest x-ray or a negative QuantiFERON test.
5. Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose.
6. History of significant other medical conditions, which in the Investigator's opinion would exclude the patient from participating in this trial.
7. History of recurrent and/or evidence of active bacterial, fungal, or viral infection(s).
8. Use of prohibited therapies, any other investigational biologics within 8 weeks prior to the Baseline visit, any other investigational drugs, other than investigational biologic treatment, within 30 days (or 3 months for investigational monoclonal antibodies) or 5 half-lives prior to the Baseline visit, whichever is longer
9. History of known hypersensitivity to canakinumab.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Galway, Ireland, Ireland
- Italy (4):
  - Novartis Investigative Site, Sciacca, AG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pavia, PV
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Torene R, Nirmala N, Obici L, Cattalini M, Tormey V, Caorsi R, Starck-Schwertz S, Letzkus M, Hartmann N, Abrams K, Lachmann H, Gattorno M. Canakinumab reverses overexpression of inflammatory response genes in tumour necrosis factor receptor-associated periodic syndrome. Ann Rheum Dis. 2017 Jan;76(1):303-309. doi: 10.1136/annrheumdis-2016-209335. Epub 2016 Jul 29. PMID 27474763
- [Derived] Gattorno M, Obici L, Cattalini M, Tormey V, Abrams K, Davis N, Speziale A, Bhansali SG, Martini A, Lachmann HJ. Canakinumab treatment for patients with active recurrent or chronic TNF receptor-associated periodic syndrome (TRAPS): an open-label, phase II study. Ann Rheum Dis. 2017 Jan;76(1):173-178. doi: 10.1136/annrheumdis-2015-209031. Epub 2016 Jun 7. PMID 27269295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in 3 countries.
Pre-assignment Details: A total of 29 participants were screened, out of which 20 were enrolled and exposed to study medication. Nine participants were considered as screening failures due to unacceptable laboratory value or test procedure results.
Groups:
- Canakinumab: Participants received body-weight stratified dosage of canakinumab (2 milligram/ kilogram (mg/kg) for participants equal to or less than (≤) 40 kg or 150 mg for participants more than (>) 40 kg) through subcutaneous (s.c.) route as the starting dose at baseline and monthly for 4 months. The dose was escalated at Day 8 if dose of canakinumab was not sufficient to resolve the qualifying TNF-receptor associated periodic syndrome (TRAPS) flare.
Period: Overall Study
Arm/Group | Canakinumab
Started | 20
Completed | 18
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The analysis was performed on Safety Set (SAF) defined as all participants who received at least one application of study treatment and had least one post-baseline safety assessment.
Groups:
- Canakinumab: Participants received body-weight stratified dosage of canakinumab (2 mg/kg for participants ≤ 40 kg or 150 mg for participants > 40 kg) through s.c. route as the starting dose at baseline and monthly for 4 months. The dose was escalated at Day 8 if dose of canakinumab was not sufficient to resolve the qualifying TRAPS flare.
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.62 (18.362)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  Ireland | 2
  Italy | 10
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete or Almost Complete Response at Day 15
Description: Complete response was defined as clinical remission and serological remission. Clinical remission was defined as Physician's Global Assessment of TRAPS activity absent or minimal and serological remission was defined as C reactive protein (CRP) and/or Serum amyloid A protein (SAA) to be less than (<) 10 milligram per liter (mg/L). Almost complete response was defined as clinical remission and a partial serological remission (equal to or more than [≥] 70% reduction of baseline CRP and/or SAA).
Time Frame: Day 15
Population: The primary analysis was performed on the Full Analysis Set (FAS), defined as all participants who received at least one dose of study treatment and had at least one post-baseline assessment for primary efficacy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants | 95 [75.1 to 99.9]

2. Secondary Outcome: Percentage of Participants With Complete or Almost Complete Response at Day 8
Description: Complete response was defined as clinical remission and serological remission. Clinical remission was defined as Physician's Global Assessment of TRAPS activity absent or minimal and serological remission was defined as CRP and/or SAA < 10 mg/L. Almost complete response was defined as clinical remission and a partial serological remission (≥70% reduction of baseline CRP and/or SAA).
Time Frame: Day 8
Population: The analysis was performed on the FAS population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants | 80 [56.3 to 94.3]

3. Secondary Outcome: Percentage of Participants With Complete Clinical Remission at Day 8 and 15
Description: Complete clinical remission was defined as Physician's Global Assessment of TRAPS activity to be absent or minimal (1). TRAPS associated clinical signs and symptoms were assessed by the investigator at every visit on a 5-point scale: 0 = Absent; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Day 8 and Day 15
Population: The analysis was performed on the FAS population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants
  Day 8 | 90 [68.3 to 98.8]
  Day 15 | 100 [83.2 to 100]

4. Secondary Outcome: Percentage of Participant With Target Levels of C-reactive Protein (CRP) and Serum Amyloid A Protein (SAA) at Day 8 and 15
Description: The CRP and SAA were used as inflammatory markers. The target level concentration was ≤ 10 mg/L.
Time Frame: Day 8 and Day 15
Population: The analysis was performed on the FAS population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants
  Day 8 | 35 [15.4 to 59.2]
  Day 15 | 60 [36.1 to 80.9]

5. Secondary Outcome: Time to Physician's Assessed Clinical Remission
Description: Time period for complete remission after initial canakinumab treatment as assessed by participants was defined as a Physician's Global Assessment of TRAPS symptoms of scale 1 or less. The physician's Global Assessment was based on a 5-point scale: 0 = None/absent ; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Baseline up to Day 15
Population: The analysis was performed on the FAS population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Days | 4 [3 to 8]

6. Secondary Outcome: Percentage of Participants With Complete or Almost Complete Response at Day 15 After Receiving Additional Dose at Day 8
Description: Participants who had not achieved a complete response at Day 8 were given an additional dose of canakinumab. Complete response was defined as clinical remission (Physician's Global Assessment of TRAPS activity absent or minimal) and serological remission (CRP and/or SAA < 10 mg/L). Almost complete response was defined as clinical remission and a partial serological remission (≥ 70% reduction of baseline CRP and/or SAA).
Time Frame: Day 15
Population: The analysis was performed on the FAS population. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 4
Percentage of participants | 100 [39.8 to 100]

7. Secondary Outcome: Time to Participant's Assessed Clinical Remission
Description: Time period for complete remission after initial canakinumab treatment as assessed by participants was defined as a participant's Global Assessment of TRAPS symptoms of scale 1 or less. The participant's Global Assessment was based on a 5-point scale: 0 = None/absent (no) ; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Baseline up to Day 15
Population: The analysis was performed on the FAS population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Days | 3 [1 to 11]

8. Secondary Outcome: Percentage Change From Baseline in C-reactive Protein (CRP) and Serum Amyloid A (SAA) Concentration to End of Study
Description: The CRP and SAA were used as inflammatory markers. The target level concentration was ≤ 10 mg/L. Negative percent change in concentration of inflammatory markers indicated improvement.
Time Frame: Day 1 up to Day 953 (End of study)
Population: The analysis was performed on the FAS population.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percent change
  CRP | -92.19 [-99 to 43.6]
  SAA | -96.54 [-99.8 to 68.3]

9. Secondary Outcome: Percentage of Participants With Defined Grades for Skin Rash, Eye Manifestations, Extremity Pain and Abdominal Pain
Description: TRAPS signs and symptoms were assessed in 4 key categories: skin disease (skin rash), eye manifestations, extremity pain (musculoskeletal), and abdominal pain. Participants were assessed for TRAPS associated signs and symptoms a 5-point Physician's global assessment scale: None/absent (no); 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Day 113 (end of treatment period) up to Day 925 (End of study)
Population: The analysis was performed on the FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants
  Skin rash absent | 95
  Skin rash minimal | 5
  Skin rash mild | 0
  Skin rash moderate | 0
  Skin rash severe | 0
  Eye manifestations absent | 90
  Eye manifestations minimal | 10
  Eye manifestations mild | 0
  Eye manifestations moderate | 0
  Eye manifestations severe | 0
  Extremity pain absent | 90
  Extremity pain minimal | 5
  Extremity pain mild | 5
  Extremity pain moderate | 0
  Extremity pain severe | 0
  Abdominal pain absent | 95
  Abdominal pain minimal | 5
  Abdominal pain mild | 0
  Abdominal pain moderate | 0
  Abdominal pain severe | 0

10. Secondary Outcome: Percentage of Participants With Defined Grades in Physician's Global Assessment Score
Description: Participants were assessed based by physician on Physician's Global Assessment measured on a 5-point scale for TRAPS associated signs and symptoms as: 0 = None/absent; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Day 1 up to Day 953 (End of study)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 18
Percentage of participants
  None | 84.2
  Minimal | 10.5
  Mild | 0
  Moderate | 0
  Severe | 0

11. Secondary Outcome: Percentage of Participants With Defined Grades in Participant's Global Assessment Score
Description: Participants assessed the disease condition based on a 5-point participant's global assessment scale based on TRAPS associated signs and symptoms as: 0 = None/absent; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Day 1 up to Day 253 (End of follow-up period)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 12
Percentage of participants
  Absent | 41.7
  Minimal | 33.3
  Mild | 8.3
  Moderate | 16.7
  Severe | 0

12. Secondary Outcome: Percentage of Relapsed Participants
Description: Relapse was defined as a Physician's Global Assessment score of 2 (and an increase of at least 1 point compared to Day 15) and CRP and/or SAA ≥ 30 mg/L representing a 30% increase from Day 15.
Time Frame: Day 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365, 393, 421, 449,477,505, 533, 561, 589, 617, 645, 673,701, 729,757, 785, 813, 841,869, 897, 925 and 953
Population: The analysis was performed on the FAS population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants
  Day 15 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 29 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 57 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 85 | 5 [0.1 to 24.9]
  Day 113 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable..
  Day 141 | 10 [1.3 to 33.1]
  Day 169 | 10 [1.9 to 45.5]
  Day 197 | 35 [30.8 to 89.1]
  Day 225 | 10 [6.8 to 93.2]
  Day 253 | 10 [1.2 to 31.7]
  Day 281 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 309 | 10 [1.2 to 31.7]
  Day 337 | 5 [0.1 to 24.9]
  Day 365 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 393 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 421 | 5 [0.1 to 27.3]
  Day 449 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 477 | 5 [0.1 to 26.0]
  Day 505 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 533 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 561 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 589 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 617 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 645 | 5 [0.5 to 71.6]
  Day 673 | 15 [3.6 to 41.4]
  Day 701 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 729 | 5 [0.1 to 27.3]
  Day 757 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 785 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 813 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 841 | 10 [1.4 to 34.7]
  Day 869 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  Day 897 | 10 [1.4 to 34.7]
  Day 925 | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.
  End of Study (Day 953) | 0 [NA to NA] — As no participant relapsed at the specified time-points, the confidence Interval value was not applicable.

13. Secondary Outcome: Time to Relapse After Last Dose of Canakinumab
Description: as for outcome 12
Time Frame: Day 85 to Day 253 (End of treatment period to Follow-up period)
Population: The analysis was performed on the FAS population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Days | 91.5 [65 to 117]

14. Secondary Outcome: Percentage of Participants Who Relapsed and Received Rescue Medication
Description: Participants who relapsed after the last dose of canakinumab and received either corticosteroid treatment or NSAID or both corticosteroid treatment and NSAID as rescue medication.
Time Frame: Day 85 to Day 953 (End of treatment period to End of study)
Population: The analysis was performed on the FAS population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Percentage of participants
  Corticosteroid | 25 [8.7 to 49.1]
  NSAID | 25 [8.7 to 49.1]
  Both corticosteroid and NSAID | 10 [1.2 to 31.7]

15. Secondary Outcome: Serum Concentration of Canakinumab
Description: Canakinumab concentrations in serum were assessed for evaluating pharmacokinetics of the drug.
Time Frame: Day 3, 8, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365, 393, 421, 449, 533, 561, 589, 617, 645, 673, 729, 785, 841, 897, 925 and 953
Population: The analysis was performed on the FAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: microgram(s)/milliliter
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
microgram(s)/milliliter
  Day 3 (n=20) | 12.737 (5.3158)
  Day 8 (n=19) | 13.874 (4.5851)
  Day 15 (n=19) | 13.609 (5.5868)
  Day 29 (n=20) | 9.911 (4.2272)
  Day 57 (n=20) | 13.605 (5.4975)
  Day 85 (n=20) | 15.291 (6.4353)
  Day 113 (n=20) | 15.837 (6.828)
  Day 141 (n=17) | 8.799 (3.1486)
  Day 169 (n=12) | 5.655 (2.2158)
  Day 197 (n=8) | 3.906 (1.6446)
  Day 225 (n=2) | 2.725 (1.2799)
  Day 253 (n=9) | 10.261 (7.9592)
  Day 281 (n=20) | 9.759 (4.6194)
  Day 309 (n=13) | 13.088 (4.6648)
  Day 337 (n=11) | 13.182 (5.464)
  Day 365 (n=9) | 15.531 (6.7944)
  Day 393 (n=2) | 20.95 (1.6263)
  Day 421 (n=2) | 20.9 (2.9698)
  Day 449 (n=17) | 17.319 (6.496)
  Day 533 (n=1) | 18.4 (NA) — As there was only 1 participant analyzed at the specified time-points, so the standard deviation value was not applicable.
  Day 561 (n=4) | 15.55 (2.2128)
  Day 589 (n=5) | 16.48 (3.8134)
  Day 617 (n=17) | 14.124 (5.8931)
  Day 645 (n=1) | 7.45 (NA) — As there was only 1 participant analyzed at the specified time-points, so the standard deviation value was not applicable.
  Day 673 (n=5) | 9.802 (4.6757)
  Day 729 (n=5) | 8.912 (3.4413)
  Day 785 (n=18) | 7.757 (2.2948)
  Day 841 (n=4) | 8.528 (2.112)
  Day 897 (n=9) | 8.157 (2.6782)
  Day 925 (n=3) | 10.527 (7.4405)
  Day 953 (n=10) | 9.56 (2.9375)

16. Secondary Outcome: Serum Concentration of Total Interleukin-1β Antibody (IL-1β)
Description: Pharmacodynamics of canakinumab was assessed by total IL-1β (sum of free and bound canakinumab) concentration, determined in serum by means of competitive Enzyme-linked immunosorbent assay (ELISA) with limit of detection at 0.25 picogram/milliliter (pg/mL).
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
pg/mL
  Day 3 (n=20) | 12.616 (20.441)
  Day 8 (n=19) | 16.811 (20.237)
  Day 15 (n=19) | 10.662 (7.6915)
  Day 29 (n=20) | 9.342 (5.1266)
  Day 57 (n=20) | 10.701 (4.5329)
  Day 85 (n=20) | 11.212 (4.1552)
  Day 113 (n=20) | 14.401 (5.491)
  Day 141 (n=17) | 10.779 (4.1092)
  Day 169 (n=12) | 10.912 (8.2431)
  Day 197 (n=8) | 30.098 (41.158)
  Day 225 (n=2) | 3.52 (0.9475)
  Day 253 (n=9) | 25.002 (28.274)
  Day 281 (n=20) | 13.722 (7.5574)
  Day 309 (n=13) | 22.478 (16.688)
  Day 337 (n=11) | 19.904 (10.789)
  Day 365 (n=9) | 16.338 (5.8318)
  Day 393 (n=2) | 27.6 (10.182)
  Day 421 (n=2) | 30.65 (12.94)
  Day 449 (n=17) | 17.723 (8.8367)
  Day 533 (n=1) | 25.2 (NA) — As there was only 1 participant analyzed at the specified time-points, so the standard deviation value was not applicable.
  Day 561 (n=4) | 15.008 (5.4952)
  Day 589 (n=5) | 16.99 (5.2212)
  Day 617 (n=17) | 14.34 (6.1663)
  Day 645 (n=1) | 16 (NA) — As there was only 1 participant analyzed at the specified time-points, so the standard deviation value was not applicable.
  Day 673 (n=5) | 15.296 (11.908)
  Day 729 (n=5) | 16.702 (12.386)
  Day 785 (n=18) | 12.698 (6.0688)
  Day 841 (n=4) | 12.478 (6.9548)
  Day 897 (n=9) | 12.331 (8.032)
  Day 925 (n=3) | 15.033 (1.7502)
  Day 953 (n=10) | 11.701 (7.9172)

17. Secondary Outcome: Number of Participants With Anti-canakinumab Antibodies at Any Visit
Description: Immunogenicity assessment included determination of anti-canakinumab (ACZ885) antibodies in serum samples using BIAcore system.
Time Frame: Day 1 up to Day 953 (End of study)
Population: The analysis was performed on the FAS population.
Measure: Number; unit: Number of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 20
Number of participants | 2

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 953 (End of study)
Description: The analysis was performed in the SAF population, defined as all participants who received at least one application of study treatment and had least one post-baseline safety assessment.
Arm/Group | Canakinumab
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=20)
Pericarditis (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 3
Chalazion (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 2
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Periorbital oedema (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 1
Chest pain (General disorders) | 3
Condition aggravated (General disorders) | 3
Fatigue (General disorders) | 7
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 10
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 3
Ear infection (Infections and infestations) | 1
Enterobiasis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 2
Haemorrhoid infection (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 12
Onychomycosis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 4
Pharyngitis streptococcal (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection viral (Infections and infestations) | 2
Viral infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 2
Blood iron decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Occult blood positive (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 11
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Presyncope (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Strangury (Renal and urinary disorders) | 1
Breast cyst (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Nasal septal operation (Surgical and medical procedures) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.